CLINICAL TRIAL: NCT02091245
Title: Phase I Trial of the Selective Inhibitor of Nuclear Export, KPT-330, in Relapsed Childhood ALL and AML.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: William Lawrence and Blanche Hughes Foundation (Other); Karyopharm Therapeutics Inc (Industry)
Responsible Party: Principal Investigator, Andrew E. Place, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-563
Record Dates: First submitted 2014-03-14; First posted 2014-03-19 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Relapsed Acute Lymphoblastic Leukemia (ALL); Refractory Acute Lymphoblastic Leukemia (ALL); Relapsed Acute Myelogenous Leukemia (AML); Refractory Acute Myelogenous Leukemia (AML); Relapsed Mixed Lineage Leukemia; Refractory Mixed Lineage Leukemia; Relapsed Biphenotypic Leukemia; Refractory Biphenotypic Leukemia; Chronic Myelogenous Leukemia (CML) in Blast Crisis
Keywords: Relapsed acute lymphoblastic leukemia (ALL); Refractory acute lymphoblastic leukemia (ALL); Relapsed acute myelogenous leukemia (AML); Refractory acute myelogenous leukemia (AML); Relapsed childhood leukemia; Relapsed mixed lineage leukemia; Refractory mixed lineage leukemia; Relapsed biphenotypic leukemia; Refractory biphenotypic leukemia; Chronic myelogenous leukemia (CML) in blast crisis
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KPT-330 (Experimental): KPT-330 will be administered twice a week on Days 1 and 3 for four weeks. Starting dose 30 mg/m2.In the dose-escalation cohort, three patients will initially be enrolled at each dose level and will be monitored for a DLT during the 28-day treatment cycle before dose escalation may occur.
  Interventions: Drug: KPT-330

INTERVENTIONS:
Drug: KPT-330
  Other Names: Selinexor

SUMMARY:
This research study involves participants who have acute lymphoblastic or acute myelogenous leukemia that has relapsed or has become resistant (or refractory) to standard therapies. This research study is evaluating a drug called KPT-330. Laboratory and other studies suggest that the study drug, KPT-330, may prevent leukemia cells from growing and may lead to the destruction of leukemia cells. It is thought that KPT-330 activates cellular processes that increase the death of leukemia cells. The main goal of this study is to evaluate the side effects of KPT-330 when it is administered to children and adolescents with relapsed or refractory leukemia.

DETAILED DESCRIPTION:
The investigators are trying to determine a safe dose of KPT-330 and will be giving participants different dose levels of the study drug. Three to six participants will receive the starting dose of the drug. If the side effects are not too severe, the next group of participants will take the study drug at a higher dose level. Up to 3 dose levels of the study drug will be tested, but once each participant has been assigned a dose level, the participant will always receive the same dose. The highest dose that people can be given safely is called the maximum tolerated dose (MTD). Once the MTD is determined, up to 10 additional participants will receive that dose to further study the drug.

Participants between the age of ≥18 months (540 days) and ≤ 21 years with relapsed (second or subsequent relapse) or refractory ALL or AML will be eligible to enroll. KPT-330 will be administered twice a week on Days 1 and 3 for four weeks (a cycle is 4 weeks). All participants will receive intrathecal chemotherapy on Day 1 of each cycle. Participants with CNS-2 disease will receive additional doses of IT chemo. Pharmacokinetic (PK) samples will be collected during Cycle 1 on Days 1-3 and 15. PK samples will be collected during Cycle 2 on Day 15. Pharmacodynamic (PD) samples will be collected during Cycle 1 on Days 1-3. PD samples will be collected during Cycle 2 on Day 15. Additional optional correlative biology sample will be collected. Participants are monitored closely for adverse events. Participants will have physical exams and blood work more than once a week during all cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patient must be ≥ 12 months (365 days) and ≤ 21 years.
* Histologically confirmed diagnosis of relapsed or refractory ALL (including Burkitt leukemia), AML, mixed lineage leukemia, biphenotypic leukemia, or chronic myelogenous leukemia (CML) in blast crisis.

  * Refractory disease defined as: Persistent disease after at least two induction cycles.
  * Relapsed disease: Second or subsequent relapse, any relapse refractory to salvage chemotherapy
* Subjects must have bone marrow with ≥ 5% blasts (M2 or M3 marrow) definitively identified either on a bone marrow aspirate or biopsy sample, as assessed by morphology, immunohistochemical studies, flow cytometry, karyotype, cytogenetic testing such as fluorescent in situ hybridization (FISH) or other molecular studies.
* Subject would not benefit from additional cytotoxic chemotherapy as determined by the treating physician.
* Patients with CNS 1 or CNS 2 disease are eligible. Patients with isolated CNS relapse or CNS 3 disease are not eligible. Please refer to Section 11.1.3 for definitions of CNS disease status and interpretation of traumatic lumbar punctures.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study and meet all of the following criteria:

  * Myelosuppressive chemotherapy: 14 days must have elapsed since the completion of myelosuppressive therapy. Individuals may have received any of the following medications within 14 days without a "wash-out" period:

    * Standard maintenance therapy (vincristine, 6MP, corticosteroids, low dose methotrexate)
    * Hydroxyurea
    * Intrathecal chemotherapy with methotrexate, hydrocortisone and/or cytarabine.
  * Radiation therapy (XRT):

    * Total Body Irradiation (TBI) or craniospinal radiation therapy: Must have been completed more than 90 days from study entry
    * Palliative XRT: XRT for chloromas does not require a washout period.
  * Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
  * Immunotherapy: At least 6 weeks after the completion of any type of immunotherapy, e.g. tumor vaccines and chimeric antigen receptor T-cells.
  * Monoclonal antibodies: At least 3 half-lives of the antibody after the last dose of a monoclonal antibody. (See table on DVL homepage listing monoclonal antibody half-lives: https://members.childrensoncologygroup.
* Performance status:

  -- Lansky ≥ 50 for individuals 18 months- ≤ 16 years old; Karnofsky > 50% for individuals 17-21 years old (See Appendix I).
* Adequate organ function defined as the following:

  * Direct bilirubin ≤1.5 X institutional upper limit of normal (ULN)
  * AST (SGOT)/ALT (SGPT) ≤ 3X institutional ULN
  * Creatinine below institutional ULN or creatinine clearance ≥ 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
  * Echocardiogram must have a shortening fraction or an ejection fraction greater than institutional lower limit of normal for age and gender. Echocardiogram must be obtained while patient is not receiving cardiotropic medications (eg., pressors or afterload reducers).
* Oxygen saturation over 90% by pulse oximetry without administration of supplemental oxygen.
* Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
* Female patients with infants must agree not to breastfeed their infants while on this study.
* The effects of KPT-330 on the developing human fetus are unknown. For this reason and because many chemotherapeutic agents are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability of participant (or parent/guardian for participants who are minors) to understand and the willingness to sign the written informed consent document.

Exclusion Criteria:Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.

* Inability to take or tolerate enteral medications
* Individuals with CNS 3 leukemia
* Individuals with Down syndrome
* Patients with prior hematopoietic stem cell transplant (HSCT) are eligible, with the exception of the following:

  * Autologous HSCT within 60 days of study entry
  * Allogeneic HSCT within 90 days of study entry
  * Evidence of graft-versus-host-disease (GVHD)
  * Treatment with immunosuppressive medications within 14 days; however, weaning or stable doses of steroids (must be ≤ 20 mg/m2/day of prednisone equivalents) and/or calcineurin inhibitors are permitted.
* Treatment with hematopoietic growth factors (G-CSF):

  * Long-acting (e.g., Neulasta) within 14 days prior to study entry
  * Short-acting (e.g., Neupogen) within 7 days prior to study entry
* Treatment with an investigational agent within 28 days of study entry, or 3 half-lives, whichever is longer.
* Patients will be excluded if there is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.
* Any ECG abnormality that in the opinion of the principal investigator would preclude safe participation in the study
* Patients refractory to red blood cell or platelet transfusions.
* Patients receiving anti-coagulation therapy are eligible as long as anti-coagulation regimen has been stable for > 1 month.
* Patients with systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment.
* For dose-escalation cohort only, known positivity for human immunodeficiency virus (HIV); baseline testing for HIV is not required. HIV positive patients will be eligible for the dose-expansion cohort.
* Known active hepatitis A, B, or C infection; or known to be positive for HCV RNA or HBsAg (HBV surface antigen); baseline testing for viral hepatitis is not required.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of KPT-330 (e.g. ulcerative colitis, uncontrolled nausea, vomiting, diarrhea, malabsorption or history of small bowel resection)
* Individuals with significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Individuals with a history of a different malignancy (other than acute leukemia) are ineligible except for the following circumstances: Individuals are eligible if the different malignancy is in complete remission at the time of study entry.
* Pregnant women are excluded from this study because KPT-330 is a chemotherapeutic agent with unknown teratogenic or abortifacient effects.
* Individuals who are eligible for allogeneic hematopoietic stem cell transplantation (HSCT) as determined by the treating physician, and have a suitable donor or appropriate stem cell source available
* Individuals who would benefit from additional cytotoxic chemotherapy as determined by the treating physician

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03; Primary Completion 2018-02 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Toxicity profile of KPT-330 assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 3 Years
  Toxicities will be tabulated by type and grade.
Maximum tolerated dose (MTD) of KPT-330 determined by incidence of dose limiting toxicities. | 2 Years
  Toxicities graded by CTCAE version 4.0

SECONDARY OUTCOMES:
Measurement of KPT-330 in the blood, urine and cerebrospinal fluid. | 2 Years
  Pharmacokinetic analysis
Assessment of anti-leukemic activity of KPT-330 measured by objective response rates. | 3 Years
Biomarker analysis including measurements of cytokine levels and expression of XPO1 in white blood cells. | 3 Years
  Pharmacodynamic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E Place, MD,PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (10):
- United States (10):
  - UCSF, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin